CLINICAL TRIAL: NCT02128815
Title: Evaluating the Effect of a Diabetes Health Coach in Individuals With Type 2 Diabetes
Acronym: DiabCoach
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: Coaching2014#
Record Dates: First submitted 2014-04-28; First posted 2014-05-01 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2017-09

CONDITIONS: Type 2 Diabetes
Keywords: adults; coaching; type 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Coaching (Experimental): diabetes health coaching + usual diabetes self-management education
  Interventions: Other: Coaching
- Usual Care (No Intervention): Usual care or self-management education

INTERVENTIONS:
Other: Coaching — Care translation - behaviour modification, personalized/tailored diabetes education and psychosocial support
  Arms: Coaching

SUMMARY:
Background: Health coaching is defined as health education, promotion and support by a professional to enhance the well-being of individuals and facilitate the achievement of their health-related goals. However, health coaching has not been adequately assessed in the community health care setting in individuals with T2DM. The purpose of this study is to determine the effect of diabetes health coaching in adults with T2DM in the community health care setting on clinical outcomes, self-care behaviours and health care utilization.

DETAILED DESCRIPTION:
Evaluating the Effect of a Diabetes Health Coach in Individuals with Type 2 Diabetes.

Background: Health coaching is defined as health education, promotion and support by a professional to enhance the well-being of individuals and facilitate the achievement of their health-related goals. However, health coaching has not been adequately assessed in the community health care setting in individuals with T2DM. The purpose of this study is to determine the effect of diabetes health coaching in adults with T2DM in the community health care setting on clinical outcomes, self-care behaviours and health care utilization.

Research Questions: In adults with T2DM who are referred to a community based diabetes program, does assignment to a diabetes health coach that provides remotely delivered frequent personalized education and support, behaviour modification counselling and reinforcement, and psychosocial support improve glycated hemoglobin (A1C) over diabetes education alone? Secondary Questions include: i) Does the assignment to a diabetes health coach improve: a) body mass index (BMI); b) diabetes self-care activities; and c) quality of life, more than standard diabetes self-management education alone after one year? ii) What is the incremental cost-effectiveness of the diabetes health coach relative to standard diabetes self-management education?

Proposed Design and Intervention:

The study design will be an open-label randomized controlled trial of adults with T2DM in a Community Health Centre (CHC) setting. Upon randomization to the intervention group, study participants will receive one-year access to diabetes health coaching, which comprises: a) weekly access to a coach, via secured messaging or telephone; b) diabetes case management; c) personalized diabetes education; d) behaviour modification, goal setting and reinforcement; and d) psychosocial support. All study participants will have access to their standard diabetes care and access to the Virtual Lifestyle Management program, an internet based deliverable program which comprises the National Institutes of Health's Diabetes Prevention Program (DPP) protocol and curriculum, proven to be effective for weight management. Education includes 24 modules with streaming audio narration; and b) tracking tools to record dietary and physical activity results. All participants will also receive an accelerometer to measure physical activity (steps).

Outcome:

The primary outcome is the difference the mean A1C in the diabetes health coaching program, compared to the mean A1C in the control group at 1 year. Secondary outcomes will include: a) BMI; b) diabetes self-care activities; c) quality of life; and d) cost-effectiveness.

Implications:

The findings from this trial may support a new strategy to complement and/or enhance diabetes self-management services in the community. Coaching may be delivered remotely and may demonstrate to be a cost-effective or cost-neutral service to support those living with diabetes.

ELIGIBILITY:
Inclusion Criteria:

* adults 18 years of age or older
* diagnosed type 2 diabetes
* A1C equal to or over 7.5%
* able to read, write and understand English
* have telephone or internet access

Exclusion Criteria:

* adults with impaired cognition
* cohabiting with a participant in the study
* pregnant or planning a pregnancy
* have an underlying medical condition that may provide misleading A1C levels

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 366 (Actual)
Dates: Start 2015-01; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
change from baseline A1C after one year | 1 year
  non-fasting venous blood sample (Hemoglobin A1C assay)

SECONDARY OUTCOMES:
BMI | change from baseline in BMI at 1 year
  The BMI is defined as the body mass divided by the square of the body height, and is universally expressed in units of kg/m2, resulting from mass in kilograms and height in metres.
Change from baseline self-care behaviours at 1 year | 1 year
  measured by the Diabetes self-care activities scale.
change from baseline in quality of life at 1 year | 1 year
  Audit of Diabetes Dependent Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Diana Sherifali, PhD, Principal Investigator — McMaster University
Locations (2):
- Canada (2):
  - Langs Community Health Centre, Cambridge, Ontario
  - McMaster University, Hamilton, Ontario

IPD SHARING:
Plan to Share IPD: Undecided
This option is still being explored.

REFERENCES:
- [Derived] Sherifali D, Brozic A, Agema P, Punthakee Z, McInnes N, O'Reilly D, Usman Ali RM, Ibrahim S, Gerstein HC. Effect of Diabetes Health Coaching on Glycemic Control and Quality of Life in Adults Living With Type 2 Diabetes: A Community-Based, Randomized, Controlled Trial. Can J Diabetes. 2021 Oct;45(7):594-600. doi: 10.1016/j.jcjd.2020.11.012. Epub 2020 Dec 5. PMID 33582039